CLINICAL TRIAL: NCT04491591
Title: Implementing Breast Reconstruction Clinical Decision Support in Diverse Practice Settings
Brief Title: Implementing BREASTChoice Into Practice
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 202005217; R18HS026699 (AHRQ)
Record Dates: First submitted 2020-07-24; First posted 2020-07-29 (Actual); Results first posted 2024-08-12 (Actual); Last update posted 2024-08-12 (Actual); Status verified 2024-08

CONDITIONS: Breast Reconstruction; Breast Cancer
Keywords: Breast cancer; Breast Reconstruction; Breast Reconstruction Education; Breast Reconstruction Decision Tool
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- BREASTChoice (Experimental): * After consent, the participant will be randomized
  * Depending on the clinic work-flow, the patient will be sent the link to the BREASTChoice tool by email or MyChart message
    * 1) prior to their visit with the surgeon;
    * 2) at the time of their visit with the surgeon;
    * 3) after the surgeon appointment
  * Will receive an online survey to complete after viewing the BREASTChoice tool assessing socio-demographics, knowledge, health literacy, decisional conflict, patient engagement, health-related quality of life, preferred decision role, and usability of the website.
  * Will pull from the electronic medical record breast cancer diagnosis stage, previous breast cancer surgery and participants' reconstruction decision after enrollment.
  Interventions: Other: Breast Reconstruction Education and Support Tool (BREASTChoice)
- Attention Control Website (Active Comparator): * After consent, the participant will be randomized
  * Depending on the clinic work-flow, the patient will be sent the link to the website by email or MyChart message
    * 1) prior to their visit with the surgeon;
    * 2) at the time of their visit with the surgeon;
    * 3) after the surgeon appointment
  * Will receive an online survey to complete after viewing the website assessing socio-demographics, knowledge, preferences, health literacy, decisional conflict, measure of patient engagement, health-related quality of life, preferred decision role, consult time, and usability of the website.
  * Will pull from the electronic medical record breast cancer diagnosis stage, previous breast cancer surgery and participants' reconstruction decision after enrollment.
  Interventions: Other: Attention Control Website
- Clinicians (Experimental): * Will receive a brief virtual training on how BREASTChoice functions and the features, including placement of the patient tool summary in the electronic health record
  * Will complete pre-post trial survey about shared decision making
  Interventions: Other: Clinician Survey

INTERVENTIONS:
Other: Breast Reconstruction Education and Support Tool (BREASTChoice) — The tool is an interactive website and can be sent through My Chart and integrated into the electronic health record
  Other Names: BREASTChoice
  Arms: BREASTChoice
Other: Attention Control Website — -(https://www.cancer.gov/types/breast/reconstruction-fact-sheet)
  Arms: Attention Control Website
Other: Clinician Survey — -Questions regarding opinions on shared decision-making with answers ranging from 1-7 with 1=strongly disagree or harmful to 7=strongly agree or beneficial. The higher the score the more the physician agrees with shared decision making.
  Arms: Clinicians

SUMMARY:
Breast reconstruction after mastectomy is a highly personal decision. Although it can restore quality of life for many, there are numerous risks associated with the procedure. The risk of complications exceeds that of most elective procedures. In past work, a clinical decision support tool, BREASTChoice, with personalized risk information and patient preferences, was created to be used to address these issues. It was modified with extensive stakeholder input and built to be incorporated into electronic health records and patient portals. This randomized control trial will evaluate whether the implementation of BREASTChoice into routine care delivery is more effective than a control website, at improving the quality of reconstruction decisions.

DETAILED DESCRIPTION:
Prior to the beginning of the Randomized Control Trial (RCT), a pilot phase will be launched to test the workflow and procedures. The investigators plan to recruit up to 20 patients, continuing until procedures are smooth and ready for the randomized trial. The investigators will follow these same procedures as the trial, other than randomization, to test the workflow and tool use programming.

For the RCT, patients considering mastectomy at academic and community practices (n=340) will be randomized over 18 months to use BREASTChoice or a control website.

After the patient participant consents to be in the study, they will be randomized (using computer random assignment) participants to view the clinical decision support tool, BREASTChoice or the attention control website, using block randomization (block size of 2 and 4). Depending on the clinic work-flow, the patients may be sent the link to the tool or control website: 1) by email or MyChart message, prior to their visit with the plastic or reconstruction surgeon, for them to complete from home or in the waiting room (ideal and preferred approach); 2) by email or MyChart, in person or virtually at the time of their plastic or reconstruction visit, for patients that have same-day breast surgeon and plastic reconstruction surgeon visits, with time to wait in between appointments; or 3) by email or MyChart, after the plastic surgery appointment, if they have not yet made a decision about reconstruction after mastectomy (e.g., if they are undergoing neoadjuvant chemotherapy, or they want or need more time to decide on their surgery choices). Participants will be sent the link via MyChart unless they do not have a MyChart account. In that case, they will be sent the link via email. Study staff will be available to answer questions about MyChart via phone or email.

BREASTChoice is interactive with multiple modules. It starts with facts about breast reconstruction. Modules describe pros and cons of reconstruction, reconstruction timing, and reconstruction types. When discussing reconstruction timing, a risk prediction model pulls health data from the EHR (asking patients information in the model that is missing) to personalize risk of complications from immediate breast reconstruction. It also shows average risks for mastectomy alone and mastectomy plus immediate breast reconstruction so women can compare their personalized risk to average risks. Each module contains real patient quotes, a section called "Let's review" which checks patients' understanding, and "What matters to you", which elicits patients' preferences. Diverse patient photos and outcomes are provided. It is written at a 7th grade reading level. Data on patients' risks and a summary of her preferences are sent to their plastic/reconstructive surgeon to view in the electronic health record. The tool takes the patient about 20minutes to complete.

Control Website: The investigators chose an attention control, rather than usual care, to reduce differences between arms in participant expectation of benefit. Those in the control arm will get a link to an NCI website about breast reconstruction. That website includes 10 sections with information about types of breast reconstruction, timing, recovery, risks, cancer surveillance and additional resources. The website provides information, but does not include values clarification or tailored risk information. It is not interactive and does not include photos..

(https://www.cancer.gov/types/breast/reconstruction-fact-sheet)

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Diagnosis of incident or recurrent stage 0-III breast carcinoma

Exclusion Criteria:

* Stage IV breast carcinoma
* Histology type besides ductal/lobular carcinoma (e.g. phyllodes, sarcoma - these rare tumors differ in treatment and prognosis)
* Prior mastectomy and are seeking delayed breast reconstruction
* No malignancy (i.e., considering mastectomy for prophylaxis only)
* Cannot give informed consent or use provided study materials due to self-reported or observed cognitive, visual, or emotional barriers

Inclusion Criteria for Clinicians:

-Clinicians who provide breast cancer care within the plastic and reconstructive surgery at Barnes Jewish Hospital, Siteman Cancer Center, Barnes Jewish West County, Christian Hospital North East, and the Stefanie Spielman Comprehensive Breast Center of OSU who provide care for patients considering breast reconstruction after mastectomy

Exclusion Criteria for Clinicians:

-Plastic and reconstructive clinicians working at other breast clinic locations, and surgeons who do provider breast reconstruction care to patients who have undergone a mastectomy due to breast cancer

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 396 (Actual)
Dates: Start 2020-11-04 (Actual); Primary Completion 2022-07-22 (Actual); Study Completion 2023-02-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mary Politi, Ph.D., Principal Investigator — Washington University School of Medicine; Clara Lee, M.D., MPP, Principal Investigator — Ohio State University
Locations (2):
- United States (2):
  - Washington University School of Medicine, St Louis, Missouri
  - The Ohio State University Wexner Medical Center, Columbus, Ohio

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | BREASTChoice | Attention Control Website | Clinicians
Started | 187 | 186 | 23
Completed | 156 | 165 | 20
Not Completed | 31 | 21 | 3
Not completed — Accidently randomized | 3 | 1 | 0
Not completed — Did not complete survey | 28 | 20 | 3

BASELINE CHARACTERISTICS:
Population: The overall number of baseline participants in the BREASTChoice arm do not include the 3 participants who were accidently randomized. The overall number of participants in the Attention Control Website arm does not include the 1 participant who was accidently randomized.
Groups:
- Total: Total of all reporting groups
Arm/Group | BREASTChoice | Attention Control Website | Clinicians | Total
Number analyzed (Participants) | 184 | 185 | 23 | 392
Age, Categorical [Count of Participants; unit: Participants] — Population: Age was not collected on Clinicians.
  Participants
    number analyzed (Participants) | 184 | 185 | 0 | 369
    <=18 years | 0 | 0 | 0 | 0
    Between 18 and 65 years | 156 | 158 | 0 | 314
    >=65 years | 28 | 27 | 0 | 55
Age, Continuous [Mean (Full Range); unit: years] — Population: Age was not collected on Clinicians.
  years
    number analyzed (Participants) | 184 | 185 | 0 | 369
    (all) | 51.0 [31 to 75] | 51.2 [25 to 75] |  | 51.3 [25 to 75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 184 | 185 | 12 | 381
  Male | 0 | 0 | 11 | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 5 | 0 | 7
  Not Hispanic or Latino | 182 | 180 | 23 | 385
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 2 | 3 | 4 | 9
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 11 | 21 | 0 | 32
  White | 167 | 156 | 19 | 342
  More than one race | 4 | 3 | 0 | 7
  Unknown or Not Reported | 0 | 2 | 0 | 2
Region of Enrollment [Number; unit: participants]
  United States | 184 | 185 | 23 | 392
Breast cancer stage [Count of Participants; unit: Participants] — * Stage IV was a criterion for exclusion, participants were included if they were eligible at the time of enrollment, but upstaged after enrollment.
  * The staging system used for breast cancer is the American Joint Committee on Cancer TNM system. The lower the stage, the less the cancer has spread. A higher stage means cancer has spread more.
  * Stage depends on the size of the cancer tumor and whether or not it has grown into nearby tissue (T), whether there is cancer in the lymph nodes (N), and whether the cancer has spread to other parts of the body beyond the breast (M). Population: This data was not collected on Clinicians.
  Participants
    Stage 0: number analyzed (Participants) | 184 | 185 | 0 | 369
    Stage 0 | 41 | 32 |  | 73
    Stage I: number analyzed (Participants) | 184 | 185 | 0 | 369
    Stage I | 75 | 77 |  | 152
    Stage II: number analyzed (Participants) | 184 | 185 | 0 | 369
    Stage II | 45 | 54 |  | 99
    Stage III: number analyzed (Participants) | 184 | 185 | 0 | 369
    Stage III | 22 | 19 |  | 41
    Stage IV: number analyzed (Participants) | 184 | 185 | 0 | 369
    Stage IV | 1 | 3 |  | 4
Annual household income [Count of Participants; unit: Participants] — There are participants excluded because they skipped the income question. Population: This data was not collected on Clinicians.
  Participants
    <$30,000: number analyzed (Participants) | 152 | 158 | 0 | 310
    <$30,000 | 12 | 17 |  | 29
    $30,000 to $74,999: number analyzed (Participants) | 152 | 158 | 0 | 310
    $30,000 to $74,999 | 33 | 28 |  | 61
    $75,000 or more: number analyzed (Participants) | 152 | 158 | 0 | 310
    $75,000 or more | 91 | 96 |  | 187
    Prefer not to answer: number analyzed (Participants) | 152 | 158 | 0 | 310
    Prefer not to answer | 16 | 17 |  | 33
Educational attainment [Count of Participants; unit: Participants]
  High school or less | 15 | 16 | 0 | 31
  Technical training | 5 | 5 | 0 | 10
  Some college | 26 | 22 | 0 | 48
  College degree | 47 | 58 | 0 | 105
  Graduate/professional degree | 49 | 57 | 23 | 129

OUTCOME MEASURES:

1. Primary Outcome: Knowledge as Measured by Decision Quality Instrument
Description: -The validated Breast Reconstruction Decision Quality Instrument (DQI) knowledge scale contains 9 items on key facts about reconstruction. A value of 1 is given for each correct answer and a value of 0 is given for each incorrect answer. An overall knowledge score is calculated for each patient by dividing the number of correct responses (range 0-9) by 9 to be re-scaled from 0-100. Higher values indicate higher knowledge.
Time Frame: After initial visit but before surgery, estimated to be before day 7
Population: Overall number of participants analyzed include those in the intent to treat analysis. Data for this outcome measure was not collected on Clinicians.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | BREASTChoice | Attention Control Website | Clinicians
Number analyzed (Participants) | 156 | 165 | 0
score on a scale | 66.7 [66.7 to 77.8] | 66.7 [55.6 to 77.8] |
Statistical Analysis 1: Comparison: BREASTChoice vs Attention Control Website; Test type: Superiority; p = 0.801, Kruskal-Wallis

2. Primary Outcome: Preference Concordance
Description: * Investigators will estimate the patient's preferred treatment (mastectomy alone vs. mastectomy with reconstruction), by inputting values (entered into BREASTChoice or control survey) into a statistical model to compute preferred treatment. The investigators will compare preferred treatments to actual treatment received, with concordance determined by agreement between preferred and actual treatment received. The investigators will consider "actual treatment received" to be delayed reconstruction, if she states an intention to have delayed reconstruction, as she might not have started this process during the study.
  * Reconstruction vs no reconstruction excluded includes those who did not have a mastectomy, unsure or no preference, or received lumpectomy.
  * Immediate vs delayed reconstruction excluded includes those with unsure preference or no preference.
  * Flap vs implant reconstruction excluded includes those unsure of final reconstruction type, unsure preference, or no preference.
Time Frame: Preference assessed after initial visit, estimated to be day 7; actual treatment received collected from the EHR
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | BREASTChoice | Attention Control Website | Clinicians
Number analyzed (Participants) | 156 | 165 | 0
Participants
  Reconstruction versus No reconstruction: Treatment matches preference | 83 | 113 |
  Reconstruction versus No reconstruction: Treatment does not match preference | 13 | 9 |
  Reconstruction versus No reconstruction: Excluded | 60 | 43 |
  Immediate reconstruction versus delayed reconstruction: number analyzed (Participants) | 103 | 109 | 0
  Immediate reconstruction versus delayed reconstruction: Treatment matches preference | 48 | 73 |
  Immediate reconstruction versus delayed reconstruction: Treatment does not match preference | 11 | 22 |
  Immediate reconstruction versus delayed reconstruction: Excluded | 44 | 14 |
  Flap reconstruction versus Implant reconstruction: number analyzed (Participants) | 103 | 109 | 0
  Flap reconstruction versus Implant reconstruction: Treatment matches preference | 33 | 60 |
  Flap reconstruction versus Implant reconstruction: Treatment does not match preference | 6 | 16 |
  Flap reconstruction versus Implant reconstruction: Excluded | 64 | 33 |
Statistical Analysis 1: Comparison: BREASTChoice vs Attention Control Website; Reconstruction versus No reconstruction; Test type: Superiority; p = 0.1336, Fisher Exact
Statistical Analysis 2: Comparison: BREASTChoice vs Attention Control Website; Test type: Superiority — Immediate reconstruction versus delayed reconstruction; p = 0.5505, Fisher Exact
Statistical Analysis 3: Comparison: BREASTChoice vs Attention Control Website; Flap reconstruction versus Implant reconstruction; Test type: Superiority; p = 0.6178, Fisher Exact

3. Primary Outcome: Decisional Conflict as Measured by the SURE (Sure of Myself; Understand Information; Risk-benefit Ratio; Encouragement) Scale for Decisional Conflict
Description: -The validated, widely-used SURE (Sure of myself; Understand information; Risk-benefit ratio; Encouragement) Measure of Decisional Conflict asks whether patients have enough information to make a choice, enough support to make a choice, and are clear about their values. It is a 4-item measure of yes/no questions (1=yes, 0=no). A score of ≤3 indicates decisional conflict; the outcome is binary indicating a score of 4 (no decisional conflict) vs. ≤3 (presence of decisional conflict).
Time Frame: After initial visit but before surgery, estimated to be before day 7
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | BREASTChoice | Attention Control Website | Clinicians
Number analyzed (Participants) | 142 | 157 | 0
Participants
  Decisional conflict | 31 | 44 |
  No decisional conflict | 111 | 113 |
Statistical Analysis 1: Comparison: BREASTChoice vs Attention Control Website; Test type: Superiority; p = 0.2317, Fisher Exact

4. Secondary Outcome: Compare Number of High-risk Participants From Each Arm Who Chose Breast Reconstruction
Description: -Participants will be considered high-risk if their risk exceeds two times the population average
Time Frame: After patient participation (approximately 18 months)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | BREASTChoice | Attention Control Website | Clinicians
Number analyzed (Participants) | 16 | 13 | 0
Participants | 10 | 11 |
Statistical Analysis 1: Comparison: BREASTChoice vs Attention Control Website; Test type: Superiority; p = 0.1052, Fisher Exact

5. Secondary Outcome: Provider Intention to Engage in Shared Decision Making as Measured by the Change in the Mean CPD (Continuing Professional Development)-Reaction Scale
Description: -The Continuing Professional Development (CPD) Reaction scale is a 12-item measure with each item having a scale of 1-7. These 12 items correspond to the following 5 constructs (2-3 items per construct) are assessed: intention (2 items), social influence (3 items), beliefs about capabilities (3 items), moral norm (2 items), and beliefs about consequence (2 items). The possible scale range is 1-7. Higher values or a positive change indicates higher intention, social influence, beliefs about capabilities, moral norm, or beliefs about consequences of engaging in shared decision making. Each scale is reported as an average.
  **For clinician arm only
Time Frame: Assessed pre- and post-study (approximately 24 months)
Population: This outcome measure is for Clinicians only.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | BREASTChoice | Attention Control Website | Clinicians
Number analyzed (Participants) | 0 | 0 | 20
score on a scale
  Intention (Pre-Study) |  |  | 6.40 (0.8)
  Intention (Post-Study): number analyzed (Participants) | 0 | 0 | 19
  Intention (Post-Study) |  |  | 6.55 (0.76)
  Social influence (Pre-Study) |  |  | 5.23 (1.78)
  Social influence (Post-Study): number analyzed (Participants) | 0 | 0 | 19
  Social influence (Post-Study) |  |  | 5.18 (1.57)
  Beliefs about capabilities (Pre-Study) |  |  | 6.04 (0.86)
  Beliefs about capabilities (Post-Study): number analyzed (Participants) | 0 | 0 | 19
  Beliefs about capabilities (Post-Study) |  |  | 6.07 (0.75)
  Moral norm (Pre-Study) |  |  | 6.43 (0.75)
  Moral norm (Post-Study): number analyzed (Participants) | 0 | 0 | 19
  Moral norm (Post-Study) |  |  | 6.68 (0.56)
  Beliefs about consequences (Pre-Study) |  |  | 6.33 (0.80)
  Beliefs about consequences (Post-Study): number analyzed (Participants) | 0 | 0 | 18
  Beliefs about consequences (Post-Study) |  |  | 6.53 (0.99)
Statistical Analysis 1: Comparison: Clinicians; Test type: Other; Within subjects pre/post comparison

6. Secondary Outcome: Knowledge as Measured by Knowledge Questions Developed in Previous Studies
Description: -This is a an 11-item measure using true/false/unsure response options. A knowledge score is calculated by dividing the number of correct responses (each scored 1 if correct, 0 if incorrect, unsure, or blank) by the number of knowledge items (11), to be re-scaled to 0-100. Higher values indicate higher knowledge.
Time Frame: After initial visit but before surgery, estimated before day 7
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | BREASTChoice | Attention Control Website | Clinicians
Number analyzed (Participants) | 156 | 165 | 0
score on a scale | 84.7 (13.8) | 66.5 (15.8) |
Statistical Analysis 1: Comparison: BREASTChoice vs Attention Control Website; Test type: Superiority; p < 0.001, Kruskal-Wallis

7. Secondary Outcome: Consult Time as Measured by Time Spent With Clinician During the Visit
Description: -Consult time using the BREASTChoice will be compared to consult using the attention control.
Time Frame: Initial visit (day 1)
Population: The data for this outcome measure was not collected.
Arm/Group | BREASTChoice | Attention Control Website | Clinicians
Number analyzed (Participants) | 0 | 0 | 0

8. Secondary Outcome: Usability as Measured by the System Usability Scale (SUS)
Description: -The System Usability Index (SUS) is a 10-item measure (each scaled 1-5) of how easy a website is to use. It is asked of only those in the BreastChoice group to assess the usability of tool. A usability score is calculated by adding the items and multiplying the sum by 2.5. Usability scores can range from 0-100 with higher scores indicating greater usability. A score greater than 68 indicates adequate usability.
Time Frame: After initial visit but before surgery, estimated to be before day 7
Population: Only participants in the BREASTChoice arm were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | BREASTChoice | Attention Control Website | Clinicians
Number analyzed (Participants) | 156 | 0 | 0
score on a scale | 84.6 (14.3) |  |
Statistical Analysis 1: Comparison: BREASTChoice; Test type: Other; Descriptive analysis using mean and standard deviation

9. Secondary Outcome: Knowledge as Measured by Decision Quality Instrument
Description: -The validated Breast Reconstruction Decision Quality Instrument (DQI) knowledge scale contains 9 items on key facts about reconstruction. A knowledge score will be calculated for each patient by dividing the number of correct responses by the number of knowledge items. Value of 1 given for each correct answer and value of 0 for each incorrect answer. Overall knowledge score range is 0-9 re-scaled from 0-100.
Time Frame: After initial visit but before surgery, estimated to be before day 7
Population: For this analysis, BREASTChoice participants who never accessed the tool were excluded. Data for this outcome measure was not collected on Clinicians.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | BREASTChoice | Attention Control Website | Clinicians
Number analyzed (Participants) | 150 | 165 | 0
score on a scale | 66.7 [66.7 to 77.8] | 66.7 [55.6 to 77.8] |
Statistical Analysis 1: Comparison: BREASTChoice vs Attention Control Website; Test type: Superiority; p = 0.0302, Kruskal-Wallis

10. Secondary Outcome: Preference Concordance as Measured by the Decision Quality Instrument
Description: * The investigators will estimate the patient's preferred treatment (mastectomy alone versus mastectomy with reconstruction), by inputting values (entered into BREASTChoice or control survey) into a statistical model to compute preferred treatment. The investigators will compare preferred treatments to actual treatment received, with concordance determined by agreement between preferred and actual treatment received. The investigators will consider "actual treatment received" to be delayed reconstruction, if she states an intention to have delayed reconstruction, as she might not have started this process during the study.
  * Reconstruction vs no reconstruction excluded includes those who did not have a mastectomy, no preference, or received lumpectomy.
  * Immediate vs delayed reconstruction excluded includes those with unsure preference or no preference.
  * Flap vs implant reconstruction excluded includes those unsure of final reconstruction type, unsure preference, or no preference.
Time Frame: Preference assessed after initial visit, estimated to be day 7; actual treatment received collected from the EHR
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | BREASTChoice | Attention Control Website | Clinicians
Number analyzed (Participants) | 150 | 165 | 0
Participants
  Reconstruction versus No reconstruction: Treatment matches preference | 83 | 113 |
  Reconstruction versus No reconstruction: Treatment does not match preference | 13 | 9 |
  Reconstruction versus No reconstruction: Excluded | 54 | 43 |
  Immediate reconstruction versus delayed reconstruction: number analyzed (Participants) | 100 | 109 | 0
  Immediate reconstruction versus delayed reconstruction: Treatment matches preference | 48 | 73 |
  Immediate reconstruction versus delayed reconstruction: Treatment does not match preference | 11 | 22 |
  Immediate reconstruction versus delayed reconstruction: Excluded | 41 | 14 |
  Flap reconstruction versus Implant reconstruction: number analyzed (Participants) | 100 | 109 | 0
  Flap reconstruction versus Implant reconstruction: Treatment matches preference | 33 | 60 |
  Flap reconstruction versus Implant reconstruction: Treatment does not match preference | 6 | 16 |
  Flap reconstruction versus Implant reconstruction: Excluded | 61 | 33 |
Statistical Analysis 1: Comparison: BREASTChoice vs Attention Control Website; Reconstruction versus No reconstruction; Test type: Superiority; p = 0.135, Fisher Exact
Statistical Analysis 2: Comparison: BREASTChoice vs Attention Control Website; Immediate reconstruction versus delayed reconstruction; Test type: Superiority; p = 0.510, Fisher Exact
Statistical Analysis 3: Comparison: BREASTChoice vs Attention Control Website; Flap reconstruction versus Implant reconstruction; Test type: Superiority; p = 0.469, Fisher Exact

11. Secondary Outcome: Decisional Conflict as Measured by the SURE (Sure of Myself; Understand Information; Risk-benefit Ratio; Encouragement) Scale for Decisional Conflict
Description: -The validated, widely-used SURE measure of decisional conflict asks whether patients have enough information to make a choice, enough support to make a choice, and are clear about their values. It is a 4-item measure of yes/no questions (1=yes, 0=no). A score of ≤3 indicates decisional conflict.
Time Frame: After initial visit but before surgery, estimated to be before day 7
Population: For this analysis, BREASTChoice participants who never accessed the tool were excluded. If participants did not answer the questions, they were also excluded. Data for this outcome measure was not collected on Clinicians.
Measure: Count of Participants; unit: Participants
Arm/Group | BREASTChoice | Attention Control Website | Clinicians
Number analyzed (Participants) | 136 | 157 | 0
Participants
  Decisional conflict | 31 | 44 |
  No decisional conflict | 105 | 113 |
Statistical Analysis 1: Comparison: BREASTChoice vs Attention Control Website; Test type: Superiority; p = 0.308, Fisher Exact

12. Secondary Outcome: Compare Number of High-risk Participants From Each Arm Who Chose Breast Reconstruction
Description: -Participants will be considered high-risk if their risk exceeds two times the population average
Time Frame: After patient participation (approximately 18 months)
Population: Only high risk participants are included in this outcome measure. Data for this outcome measure was not collected on Clinicians.
Measure: Count of Participants; unit: Participants
Arm/Group | BREASTChoice | Attention Control Website | Clinicians
Number analyzed (Participants) | 13 | 13 | 0
Participants | 8 | 11 |
Statistical Analysis 1: Comparison: BREASTChoice vs Attention Control Website; Test type: Superiority; p = 0.036, Fisher Exact

ADVERSE EVENTS:
Time Frame: Adverse events and all-cause mortality were collected through study completion (an average of 18 months).
Description: Adverse events and all-cause mortality were not collected on Clinicians.
Arm/Group | BREASTChoice | Attention Control Website | Clinicians
All-Cause Mortality (participants affected / at risk) | 0/156 | 1/165 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/156 | 0/165 | 0/0
Other Adverse Events (participants affected / at risk) | 0/156 | 0/165 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-01-20): https://cdn.clinicaltrials.gov/large-docs/91/NCT04491591/Prot_SAP_000.pdf
  • Informed Consent Form (2023-01-20): https://cdn.clinicaltrials.gov/large-docs/91/NCT04491591/ICF_001.pdf